CLINICAL TRIAL: NCT03405701
Title: The Effectiveness and Safety of in Vitro Maturation of Oocytes Versus in Vitro Fertilization in Women With High Antral Follicle Count (AFC): a Randomised Controlled Trial
Brief Title: IVM Versus IVF in High Antral Follicle Count Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS/MD/17/11
Record Dates: First submitted 2017-12-16; First posted 2018-01-23 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2018-11

CONDITIONS: PCOS; IVF; IVM

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVM (in vitro maturation) (Active Comparator): Receiving FSH (Menopur, Ferring) for 2 days on day 2/3 of the menstrual cycle (spontaneous/ OCP administration) and an ultrasound scan will be performed subsequently. Oocytes retrieval will be performed 42 hours after the last injection. Pre-maturation will last for 24-30 hours. ICSI will be used for insemination. Freeze-only on day 3 and frozen embryo transfer will be performed on the subsequent cycle using HRT protocol with a maximum of 2 embryos transferred
  Interventions: Procedure: IVM
- IVF (in vitro fertilization) (Active Comparator): Undergoing controlled ovarian hyperstimulation for in vitro Fertilization (IVF) with recombinant FSH (Menopur, Ferring) in GnRH antagonist protocol, treatment monitoring using ultrasound scans and blood tests. GnRH agonist triggering will be used for final oocytes maturation. ICSI will be used for insemination. Freeze-only on day 3 and frozen embryo transfer will be performed on the subsequent cycle using HRT protocol with a maximum of 2 embryos transferred.
  Interventions: Procedure: IVF

INTERVENTIONS:
Procedure: IVM — Patients in IVM group will receive FSH (Menopur, Ferring) for 2 days on day 2/3 of the menstrual cycle (spontaneous/ OCP administration) and the ultrasound scan will be performed subsequently. Oocytes retrieval will be performed 42 hours after the last injection. Pre-maturation will last for 24-30 hours. ICSI will be used for insemination. Freeze-only on day 3 and frozen embryo transfer will be performed on the subsequent cycle using HRT protocol with a maximum of 2 embryos transferred.
  Arms: IVM (in vitro maturation)
Procedure: IVF — Patients in IVF arm will undergo controlled ovarian hyperstimulation with recombinant FSH (Menopur, Ferring) in GnRH antagonist protocol, treatment monitoring using ultrasound scans and blood tests. GnRH agonist will be used for final oocytes maturation. ICSI will be used for insemination. Freeze-only on day 3 and frozen embryo transfer will be performed on the subsequent cycle using HRT protocol with a maximum of 2 embryos transferred.
  Arms: IVF (in vitro fertilization)

SUMMARY:
In vitro maturation (IVM) is postulated to be an alternative to conventional in vitro fertilization (IVF) to avoid ovarian hyperstimulation syndrome. This has particular potential in women with Polycystic Ovarian Syndrome (PCOS), who are at increased risk for the ovarian hyperstimulation syndrome. However, no randomized controlled trials on the comparison of IVM and conventional IVF in women with PCOS have been reported with respect to pregnancy rate and hyper-stimulation. Investigators aim to compare the effectiveness and safety of IVM with controlled ovarian hyperstimulation/IVF in women with high antral follicle count.

DETAILED DESCRIPTION:
Women with PCOS and PCOM or high AFC: ≥24 Antral Follicles in Both Ovaries will be given the information about the study during the first consultation which is at least 2 weeks before having periods. On the second day of periods, women will be screened for eligibility by the treating clinicians. Women who met the inclusion criteria will be invited to participate in the study. Women will be randomized (1:1) to IVM or IVF- GnRH agonist triggering cycle using block randomization by an independent study coordinator via telephone, using a computer-generated random list (block size 2, 4, 6 or 8).

Group 1: IVM Patients with a normal cycle length (>/=35 days) will receive injected highly purified human menopausal gonadotropin (hp-hMG; Menopur, Ferring) 150 IU/day starting on day two or three of the spontaneous menstrual cycle. Oocyte retrieval will be performed 42 hours after the last hp-hMG injection. Women who do not have a normal cycle length (>35 days; 4-9 menstrual cycles in a year or amenorrhea) will take an oral contraceptive for 2 weeks, then receive hp-hMG 150 IU/day (hp-hMG; Menopur, Ferring injection for 2 days starting 5 days later.

In all patients, ultrasound will be performed on the second day of gonadotrophin injection and OPU is scheduled for 42 hours after the last gonadotrophin injection. After oocyte pick-up, all oocytes will be placed in pre-maturation medium (CAPA Pre-maturation in Medicult IVM medium, Origio, Denmark) for 24 hours, then transferred to maturation culture (Medicult IVM system with phenol red, Origio, Denmark) for 30 hours.

Group 2: IVF All women in this group will undergo COH using a hp-hMG/GnRH antagonist protocol, with an hp-hMG dose of 150-225 IU/day (Menopur, Ferring), depending on age and body mass index. Follicular development will be monitored using ultrasound scanning, and estradiol and progesterone levels. When at least two leading follicles reach 17 mm in diameter, GnRH agonist (GnRHa) triggering with triptorelin 0.2 mg (Diphereline, Ipsen Beaufour) will be administered, and oocyte retrieval performed 36 hours later.

Laboratory procedures For both groups, insemination will be performed using intra-cytoplasmic sperm injection (3-4 hours after oocyte retrieval or maturation check); only matured oocytes will be inseminated. Fertilization check will be performed under an inverted microscope at 16-18 hours after insemination. Embryo evaluation will be performed at 68 ±1 hours after fertilization using the Istanbul consensus.

Freeze-all and Frozen embryo transfer In both groups, all embryos will be frozen on day 3. Frozen transfer of a maximum of 2 embryos will be performed in a subsequent cycle using HRT for endometrial preparation.

In the following cycle, the endometrium will be prepared using oral estradiol valerate (Valiera®; Laboratories Recalcine) 8 mg/day starting from the second or third day of the menstrual cycle. Endometrial thickness will be monitored from day six onwards, and vaginal progesterone (Cyclogest®; Actavis) 800 mg/day will be started when endometrial thickness reached 8 mm or more. A maximum of 2 embryos will be thawed on the day of embryo transfer, three days after the start of progesterone. Two hours after thawing, surviving embryos will be transferred into the uterus under ultrasound guidance. When women had more than two embryos frozen, the procedure will be repeated in subsequent cycles if they fail the first transfer.

ELIGIBILITY:
Inclusion Criteria:

* Women with high AFC (≥24 Antral Follicles in Both Ovaries), including PCOS plus PCO or high AFC
* Having indications for ART
* Having ≤ 2 IVM/IVF attempts
* Permanent resident in Vietnam
* Agree to have all embryos frozen on day 3
* Agree to have ≤ 2 embryos transferred in a subsequent frozen transfer
* Not participating in another IVF study at the same time

Exclusion Criteria:

* Oocyte donation cycles
* Pre-implantation genetic diagnosis (PGD) cycles

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 546 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Live birth after the first embryo transfer of the started treatment cycle | 12 weeks of gestation
  Live birth is defined as the birth of at least one newborn after 24 weeks' gestation that exhibits any sign of life (twins will be a single count). To allow assessment of the timing of live birth, the rate of ongoing pregnancy at 12 weeks will be used in calculations, conditional on the fact that this ongoing pregnancy results in live birth.

SECONDARY OUTCOMES:
Positive pregnancy test | at 2 weeks after the embryo placement after the completion of the first transfer
  Serum human chorionic gonadotropin level greater than 5 mIU/mL
Clinical pregnancy | 5 weeks after embryo placement after the completion of the first transfer
  at least one gestational sac on ultrasound at 7 weeks' gestation with the detection of heart beat activity
Ongoing pregnancy | at 10 weeks or beyond after the embryo placement after the completion of the first transfer
  Pregnancy with detectable heart rate at 12 weeks' gestation or beyond
Implantation rate | 3 weeks after embryo transferred after the completion of the first transfer
  as the number of gestational sacs per number of embryos transferred
Number of top quality embryos | 3 days after oocytes pick-up day in IVF or 5 days in IVM
  Top quality embryos are defined followed Istanbul consensus
Number of freezable embryos | 3 days after oocytes pick-up day in IVF or 5 days in IVM after the completion of the first transfer
  Number of frozen embryos
Time from randomisation to ongoing pregnancy | 12 weeks of gestation after the completion of the first transfer
  Time from randomization to ongoing pregnancy after the completion
Cumulative ongoing pregnancy at 6 months | at 6 months after randomization
  After 6 months, most patients doing IVM have finished all their frozen embryos. If they still fail, they usually change to IVF. We lose the comparison; therefore, we consider this time point for analyzing the cumulative ongoing pregnancy rate.
Cumulative ongoing pregnancy at 12 months | at 12 months after randomization
  After 12 months, most patients doing IVF have finished all their frozen embryos; therefore, we consider this time point for analyzing the cumulative ongoing pregnancy rate.

OTHER OUTCOMES:
Ovarian hyperstimulation syndrome (OHSS) | at 03 days after oocytes pick-up and 14 days after embryo transfer
  Routine assessments for OHSS were performed on day 3 post oocyte retrieval in both groups. At other times, OHSS was evaluated if symptoms were reported by the patient. OHSS was classified using the flow diagram developed by Humaidan and colleagues for use in clinical trial settings
Ectopic pregnancy | at 12 weeks of gestation after the completion of the first transfer
  a pregnancy in which implantation takes place outside the uterine cavity after the completion of the first transfer
Ectopic pregnancy | at 6 months after randomisation
  A pregnancy in which implantation takes place outside the uterine cavity
Ectopic pregnancy | at 12 months after randomisation
  A pregnancy in which implantation takes place outside the uterine cavity
Miscarriage | at 24 weeks of gestation after the completion of the first transfer
  pregnancy loss at < 12 weeks
Miscarriage | At 6 months after randomisation
  pregnancy loss at < 12 weeks
Miscarriage | at 12 months after randomisation
  pregnancy loss at < 12 weeks
Hypertensive disorders of pregnancy | at 20 weeks of gestation or beyond after the completion of the first transfer
  Pregnancy-induced hypertension, pre-eclampsia and eclampsia
Hypertensive disorders of pregnancy | at 20 weeks of gestation or beyond at 6 months after randomisation
  Pregnancy-induced hypertension, pre-eclampsia and eclampsia
Hypertensive disorders of pregnancy | at 20 weeks of gestation or beyond at 12 months after randomisation
  Pregnancy-induced hypertension, pre-eclampsia and eclampsia
Gestational diabetes mellitus | at 24 weeks of gestation after the completion of the first transfer
  using a 75g oral glucose tolerance test
Gestational diabetes mellitus | at 24 weeks of gestation at 6 months after randomisation
  using a 75g oral glucose tolerance test
Gestational diabetes mellitus | at 24 weeks of gestation at 12 months after randomisation
  using a 75g oral glucose tolerance test
Preterm delivery | at 24, 28, 32 weeks and 37 weeks of gestation after the completion of the first transfer
  Multiple definitions, defined as delivery at <24, <28, <32, <37 completed weeks
Preterm delivery | at 24, 28, 32 weeks and 37 weeks of gestation at 6 months after randomisation
  Multiple definitions, defined as delivery at <24, <28, <32, <37 completed weeks
Preterm delivery | at 24, 28, 32 weeks and 37 weeks of gestation at 12 months after randomisation
  Multiple definitions, defined as delivery at <24, <28, <32, <37 completed weeks
Multiple pregnancy | after the completion of the first transfer
  Defined as presence of more than one sac at early pregnancy ultrasound (6-8 weeks gestation)
Multiple pregnancy | at 6 months after randomisation
  Defined as presence of more than one sac at early pregnancy ultrasound (6-8 weeks gestation)
Multiple pregnancy | at 12 months after randomisation
  Defined as presence of more than one sac at early pregnancy ultrasound (6-8 weeks gestation)
Multiple delivery | 22 weeks of gestation or beyond after the completion of the first transfer
  Birth of more than one baby beyond 24 weeks
Multiple delivery | 22 weeks of gestation or beyond at 6 months after randomisation
  Birth of more than one baby beyond 24 weeks
Multiple delivery | 22 weeks of gestation or beyond at 12 months after randomisation
  Birth of more than one baby beyond 24 weeks
Antepartum haemorrhage | After the completion of the first transfer
  Including placenta previa, placenta accreta and unexplained
Antepartum haemorrhage | At 6 months after randomisation
  Including placenta previa, placenta accreta and unexplained
Antepartum haemorrhage | At 12 months after randomisation
  Including placenta previa, placenta accreta and unexplained
Spontaneous preterm birth | at 24, 28, 32 weeks and 37 weeks of gestation after the completion of the first transfer
  Defined as delivery at <24, <28, <32, <37 completed weeks
Spontaneous preterm birth | at 24, 28, 32 weeks and 37 weeks of gestation at 6 months after randomisation
  Defined as delivery at <24, <28, <32, <37 completed weeks
Spontaneous preterm birth | at 24, 28, 32 weeks and 37 weeks of gestation at 12 months after randomisation
  Defined as delivery at <24, <28, <32, <37 completed weeks
Iatrogenic preterm birth | at 24, 28, 32 weeks and 37 weeks of gestation after the completion of the first transfer
  Defined as delivery at <24, <28, <32, <37 completed weeks
Iatrogenic preterm birth | at 24, 28, 32 weeks and 37 weeks of gestation at 6 months after randomisation
  Defined as delivery at <24, <28, <32, <37 completed weeks
Iatrogenic preterm birth | at 24, 28, 32 weeks and 37 weeks of gestation at 12 months after randomisation
  Defined as delivery at <24, <28, <32, <37 completed weeks
Birth weight | at the time of delivery
  Weight of singletons and twins
Large for gestational age | at the time of delivery after the completion of the first transfer
  birth weight >90th percentile
Large for gestational age | at the time of delivery at 6 months after randomisation
  birth weight >90th percentile
Large for gestational age | at the time of delivery at 12 months after randomisation
  birth weight >90th percentile
Small for gestational age | at the time of delivery after the completion of the first transfer
  birth weight < 10th percentile
Small for gestational age | at the time of delivery at 6 months after randomisation
  birth weight < 10th percentile
Small for gestational age | at the time of delivery at 12 months after randomisation
  birth weight < 10th percentile
Low birth weight | at birth after the completion of the first transfer
  Weight < 2500 gm at birth
Low birth weight | at 6 months after randomisation
  Weight < 2500 gm at birth
Low birth weight | at 12 months after randomisation
  Weight < 2500 gm at birth
Very low birth weight | at birth after the completion of the first transfer
  Weight < 1500 gm at birth
Very low birth weight | at 6 months after randomisation
  Weight < 1500 gm at birth
Very low birth weight | at 12 months after randomisation
  Weight < 1500 gm at birth
High birth weight | at birth after the completion of the first transfer
  Weight >4000 gm at birth
High birth weight | at 6 months after randomisation
  Weight >4000 gm at birth
High birth weight | at 12 months after randomisation
  Weight >4000 gm at birth
Very high birth weight | at birth after the completion of the first transfer
  Weight >4500 gm at birth
Very high birth weight | at 6 months after randomisation
  Weight >4500 gm at birth
Very high birth weight | at 12 months after randomisation
  Weight >4500 gm at birth
Congenital anomaly | At 6 months after randomisation
  Any congenital anomaly will be included
Congenital anomaly | At birth after the completion of the first transfer
  Any congenital anomaly will be included
Congenital anomaly | At 12 months after randomisation
  Any congenital anomaly will be included
Admission to NICU | 7 days after delivery after the completion of the first transfer
  The admittance of the newborn to NICU
Admission to NICU | At 6 months after randomisation
  The admittance of the newborn to NICU
Admission to NICU | At 12 months after randomisation
  The admittance of the newborn to NICU
Genetic and epigenetic analysis of newborn | 1 day (Prior to the initiation of IVF/IVM) and 1 day ( at the time of delivery)
  Maternal whole blood; newborn's materials including cord blood, neonatal buccal smear, and placental tissue will be collected
Cost-effectiveness | Two year after randomization
  Including direct and indirect costs; costs related to complications treatment. Cost data will be collected for a supplementary analysis and will be reported in a separated paper.

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, MD,PhD, Principal Investigator — Mỹ Đức Hospital
Locations (1):
- Mỹ Đức Hospital, Ho Chi Minh City, Tan Binh, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saucedo-Cuevas L, Ma MPQ, Le AH, Akin N, Pham TD, Ho TM, Pita G, Gonzalez-Neira A, De Vos M, Smitz J, Anckaert E, Vuong LN. Epigenetic variation in neonatal tissues in infants conceived using capacitation-in vitro maturation vs. in vitro fertilization. Fertil Steril. 2024 Mar;121(3):506-518. doi: 10.1016/j.fertnstert.2023.11.040. Epub 2023 Dec 3. PMID 38052376
- [Derived] Vuong LN, Ho VNA, Ho TM, Dang VQ, Phung TH, Giang NH, Le AH, Pham TD, Wang R, Smitz J, Gilchrist RB, Norman RJ, Mol BW. In-vitro maturation of oocytes versus conventional IVF in women with infertility and a high antral follicle count: a randomized non-inferiority controlled trial. Hum Reprod. 2020 Nov 1;35(11):2537-2547. doi: 10.1093/humrep/deaa240. PMID 32974672
- [Derived] Vuong LN, Ho VNA, Ho TM, Dang VQ, Phung TH, Giang NH, Le AH, Pham TD, Wang R, Norman RJ, Smitz J, Gilchrist RB, Mol BW. Effectiveness and safety of in vitro maturation of oocytes versus in vitro fertilisation in women with high antral follicle count: study protocol for a randomised controlled trial. BMJ Open. 2018 Dec 9;8(12):e023413. doi: 10.1136/bmjopen-2018-023413. PMID 30530584